CLINICAL TRIAL: NCT03521505
Title: Dexmedetomidine and Brain Perfusion Monitor for Sedation of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration
Brief Title: Dexmedetomidine for Sedation of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ting-Yu Lin, Medical doctor, Assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201601093A3
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Bronchoscopy
Keywords: Sedation; dexmedetomidine; brain perfusion; bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine arm (Experimental): Dexmedetomidine will be administrated for sedation of EBUS-TBNA
  Interventions: Drug: Dexmedetomidine arm
- Propofol arm (Active Comparator): Propofol will be administrated for sedation of EBUS-TBNA
  Interventions: Drug: Propofol arm

INTERVENTIONS:
Drug: Dexmedetomidine arm — Induction: Dexmedetomidine 1ug/kg infusion for 10 minutes. 5 mg/kg alfentanil (1:10 dilution) slow injection 2 min before complete Dexmedetomidine induction Maintenance: Dexmedetomidine 0.5~1.4ug/kg/hour infusion±0.2ug/kg/hour to maintain stable vital signs and The Observer Assessment of Alertness and Sedation scale (OAA/S) 3~2. the infusion rate was increased by 0.2ug/kg/hour if the patient persistently had eye opening, talked, or became irritable and interfered with the procedure. The infusion rate was reduced by 0.2ug/kg/hour, if the following adverse events occurred: hypoxemia (SpO2 < 90%) or hypotension (mean arterial pressure (MAP) < 65 mmHg, or systolic blood pressure (SBP) < 90 mmHg) in any duration
  Arms: Dexmedetomidine arm
Drug: Propofol arm — 5 mg/kg alfentanil (1:10 dilution) slow injection 2 min before induction Induction: The initial effect-site concentration (Ce) of propofol was targeted to 2.0 μg/ml for induction (Schneider model of target-controlled infusion (TCI), Injectomat total intravenous anaesthesia (TIVA) Agilia, Fresenius Kabi, France). If OAA/S did not reach 3 while Ce achieved 2.0 μg/ml, Ce was increased by 0.2 μg/ml every 90 seconds until OAA/S 3~2.
  Maintenance: the Ce was increased by 2.0 μg/mL every 90 seconds if the patient persistently had eye opening, talked, or became irritable and interfered with the procedure. The Ce was reduced by 0.2 μg/ml every 90 seconds, if the following adverse events occurred: hypoxemia (SpO2 < 90%) or hypotension (mean arterial pressure (MAP) < 65 mmHg, or systolic blood pressure (SBP) < 90 mmHg) in any duration.
  Arms: Propofol arm

SUMMARY:
Preventing hypoxemia is one of the major goal of studies for bronchoscopic sedation. Dexmedetomidine is a sedative agents via α2 adrenergic agonist, with little respiratory suppression. In the preset study, we evaluate the safety and feasibility of the Dexmedetomidine in the specific bronchoscopic procedure, endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration.

DETAILED DESCRIPTION:
Patients undergoing flexible bronchoscopy (FB) experience procedure-related symptoms. Current guidelines of FB recommend sedation to all patients undergoing FB, except when there are contraindications. Propofol plus an opioid is the common combination used to improve patient tolerance and satisfaction during FB. However, controversy about combining propofol and opioids persists because of the risk of over-sedation and cardiopulmonary depression, especially for the time-consuming endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration (TBNA). Similar with other published data, around 40% of hypoxemia event was observed during FB sedation in the investigators' hospital. Dexmedetomidine, is a sedative agents via α2 adrenergic agonist, with little respiratory suppression. It has been applied in patients with mechanical ventilation, undergoing gastroendoscopy and extracorporal shockwave lithotripsy. Little evidences are available for Dexmedetomidine in sedation for EBUS-TBNA.

In this study, the investigators will evaluate the safety and feasibility of Dexmedetomidine for sedation of EBUS-TBNA comparing to Propofol for sedation of EBUS-TBNA. Generally, the FB sedation can divided into three parts: the induction (from starting sedative administration to insertion of bronchoscope); the maintenance ( from insertion of bronchoscope to its removal) and the recovery (from bronchoscope removal to patients gain consciousness). The primary endpoint is the proportion of patients with hypoxemia during maintenance of sedation. the investigators will also observe the other sedative outcomes, e.g. blood pressure, sedative drug dosing and patient tolerance and cooperation. The present study will also observe the association between brain perfusion and sedative outcomes via non-invasive monitor. Based on the unique pharmacokinetic property of Dexmedetomidine and the real-time brain perfusion monitor, Dexmedetomidine-based sedation may provide better safety profile for EBUS-TBNA than propofol and discover novel connection between sedative outcomes and brain perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective bronchoscopy and sedation

Exclusion Criteria:

* Age less than 20 years
* American Society of Anaesthesiologists (ASA) physical status classification IV or V
* Mallampati score of 4
* Severe sleep apnoea syndrome (apnoea-hypopnea index more than 40)
* Body mass index more than 42 in males or 35 in females
* Neurologic disorders or other conditions contributing to difficulty in assessing response
* Forced expiratory vital capacity (FVC) less than 15 ml/kg body weight, forced expiratory volume in one second (FEV1) less than 1000 ml, or FEV1/FVC less than 35%
* History of second or third degree atrioventricular block, heat rate less than 50 beat per minute or systolic blood pressure less than 90 mmHg
* Pregnancy
* Patients with a known history of allergy to the study drugs, or to eggs, soybeans or sulfite products

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin TY, Lo YL, Hsieh CH, Ni YL, Wang TY, Lin HC, Wang CH, Yu CT, Kuo HP. The potential regimen of target-controlled infusion of propofol in flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2013 Apr 24;8(4):e62744. doi: 10.1371/journal.pone.0062744. Print 2013. PMID 23638141
- [Background] Lo YL, Lin TY, Fang YF, Wang TY, Chen HC, Chou CL, Chung FT, Kuo CH, Feng PH, Liu CY, Kuo HP. Feasibility of bispectral index-guided propofol infusion for flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2011;6(11):e27769. doi: 10.1371/journal.pone.0027769. Epub 2011 Nov 23. PMID 22132138
- [Background] Lin TY, Fang YF, Huang SH, Wang TY, Kuo CH, Wu HT, Kuo HP, Lo YL. Capnography monitoring the hypoventilation during the induction of bronchoscopic sedation: A randomized controlled trial. Sci Rep. 2017 Aug 17;7(1):8685. doi: 10.1038/s41598-017-09082-8. PMID 28819181
- [Background] Ryu JH, Lee SW, Lee JH, Lee EH, Do SH, Kim CS. Randomized double-blind study of remifentanil and dexmedetomidine for flexible bronchoscopy. Br J Anaesth. 2012 Mar;108(3):503-11. doi: 10.1093/bja/aer400. Epub 2011 Dec 15. PMID 22174346
- [Result] Lin TY, Huang YC, Kuo CH, Chung FT, Lin YT, Wang TY, Lin SM, Lo YL. Dexmedetomidine sedation for endobronchial ultrasound-guided transbronchial needle aspiration, a randomised controlled trial. ERJ Open Res. 2020 Nov 10;6(4):00064-2020. doi: 10.1183/23120541.00064-2020. eCollection 2020 Oct. PMID 33693047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from chest physicians referral at a medical center between and . The first participant was enrolled in May 2018 and the last participant was enrolled in January 2020.
Pre-assignment Details: 50 subjects met inclusion criteria and were randomized to treatment.
Groups:
- Propofol Arm: Propofol will be administrated for sedation of EBUS-TBNA
  Propofol arm: 5 mg/kg alfentanil (1:10 dilution) slow injection 2 min before induction Induction: The initial effect-site concentration (Ce) of propofol was targeted to 2.0 μg/ml for induction (Schneider model of target-controlled infusion (TCI), Injectomat total intravenous anaesthesia (TIVA) Agilia, Fresenius Kabi, France). If OAA/S did not reach 3 while Ce achieved 2.0 μg/ml, Ce was increased by 0.2 μg/ml every 90 seconds until OAA/S 3~2.
  Maintenance: the Ce was increased by 2.0 μg/mL every 90 seconds if the patient persistently had eye opening, talked, or became irritable and interfered with the procedure. The Ce was reduced by 0.2 μg/ml every 90 seconds, if the following adverse events occurred: hypoxemia (SpO2 < 90%) or hypotension (mean arterial pressure (MAP) < 65 mmHg, or systolic blood pressure (SBP) < 90 mmHg) in any duration.
Period: Overall Study
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Arm | Propofol Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (14.1) | 59.4 (12.2) | 59.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25 | 25 | 50
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (3.9) | 23.6 (3.8) | 23.6 (3.8)
American Society of Anaesthesiologists physical status [Median (Full Range); unit: units on a scale] — The American Society of Anesthesiologists physical status classification system is a grading system for assessing the fitness of patients before surgery.
  A sixth category was later added. The higher grade, the poor physical status.
  1. Normal healthy patient;
  2. Patients with mild systemic disease
  3. Patients with severe systemic disease
  4. Patients with severe systemic disease that is a constant threat to life
  5. Moribund patients who are not expected to survive without the operation
  6. A declared brain-dead patient who organs are being removed for donor purposes
  units on a scale | 3 [1 to 3] | 3 [1 to 3] | 3 [1 to 3]
Mallampati score [Median (Full Range); unit: units on a scale] — Mallampati score comprises a visual assessment of the distance from the tongue base to the roof of the mouth, and therefore the amount of space in which there is to work. There are 4 scores. The higher score represents narrower space of upper airway.
  Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible.
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Hypoxemia During Maintenance
Description: The percentage of patients with hypoxemia (oxyhemoglobin saturation (SpO2)<90%) during maintenance of Bronchoscopic sedation
Time Frame: After starting bronchoscopy, up to 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
Participants | 8 | 14

2. Secondary Outcome: Hypoxemia During Induction
Description: The percentage of patients with hypoxemia (oxyhemoglobin saturation (SpO2)<90%) during induction of bronchoscopic sedation
Time Frame: After starting induction, up to 30 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
Participants | 1 | 2

3. Secondary Outcome: The Global Tolerance for Bronchoscopy
Description: The Global Tolerance of patients for bronchoscopy will be evaluated by 100-mm visual analogue scale (VAS, 0: no bother, 100: worst intolerable) after recovery
Time Frame: After recovery from sedation, up to 120 minutes
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
units on a scale | 12.5 [0 to 96] | 0 [0 to 12]

4. Secondary Outcome: The Cooperation of Patients From the View of Bronchoscopists
Description: The Cooperation of Patients will be evaluated by 100-mm visual analogue scale (VAS, 0: well cooperation, 100: worst cooperation) after recovery.
Time Frame: After recovery from sedation, up to 120 minutes
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
units on a scale | 14 [0 to 87] | 31 [1 to 70]

5. Secondary Outcome: Hypotension During Bronchoscopic Sedation
Description: The percentage of patients with hypotension (mean arterial blood pressure (MAP) less than 65 mmHg with any duration.
Time Frame: After starting sedation, up to 120 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
Participants | 1 | 5

6. Secondary Outcome: Bradycardia During Bronchoscopic Sedation
Description: The percentage of patients with bradycardia (heat beat per minute less than 60)
Time Frame: After starting sedation, up to 120 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
Participants | 12 | 4

7. Secondary Outcome: Procedure Time and Recovery Time
Description: The procedure time of bronchoscopy and recovery time from sedation to awake.
Time Frame: After starting bronchoscopy, up to 120 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine Arm | Propofol Arm
Number analyzed (Participants) | 25 | 25
minutes | 30.0 (13.2) | 27.6 (8.6)

ADVERSE EVENTS:
Time Frame: After subjects recovered from sedation, up to 30 minutes.
Arm/Group | Dexmedetomidine Arm | Propofol Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 9/25 | 17/25
Other Adverse Events (participants affected / at risk) | 16/25 | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Arm (N=25) | Propofol Arm (N=25)
Hypotension (Cardiac disorders) | 1 (1) | 5 (5)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Arm (N=25) | Propofol Arm (N=25)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 16 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Nausia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03521505/Prot_SAP_001.pdf